CLINICAL TRIAL: NCT03096899
Title: An Observational Study to Estimate Overall Survival in Patients Receiving Best Supportive Care for Treatment-Resistant, Metastatic Colorectal Carcinoma
Brief Title: A Study to Estimate Overall Survival in Patients Receiving Best Supportive Care for Treatment-Resistant, Metastatic Colorectal Carcinoma
Status: Withdrawn | Type: Observational
Why Stopped: The investigator conducting the study determined that the entry criteria for the proposed subjects was too difficult to determine in a retrospective review.
Sponsor: The Rogosin Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RI-CR-002
Record Dates: First submitted 2017-03-16; First posted 2017-03-30 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Metastatic Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — Best Supportive Care

SUMMARY:
The primary objective of this study is to estimate overall survival in patients only receiving best supportive care (BSC) for treatment-resistant, metastatic colorectal carcinoma. The primary efficacy outcome is overall survival, defined as the time from the date of the radiographic scan demonstrating disease progression post available treatments (time of origin, T0) to death from any cause.

DETAILED DESCRIPTION:
This is a retrospective chart review and prospective observational study. Patients will be considered for enrollment if they are receiving BSC and have already decided independently of this study not to pursue further therapeutic treatment of their cancer. Patients must have received at least two prior treatments for their disease, such as chemotherapy, targeted therapy or other regimens.

The study will consist of administration of informed consent, which will include permission to review medical records and record relevant medical information, agreement to be followed for survival, and evaluation of the appropriate inclusion/exclusion entry criteria.

Patients will not have any study-specific assessments performed as part of this study, and will be followed only for survival.

Approximately 80 patients with treatment-resistant, metastatic colorectal cancer who are only receiving BSC, will be entered in the study at no more than five sites in the United States

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be considered eligible to participate in the study:

1. Adult men or women, aged 18 years or older, with histologically-confirmed, metastatic adenocarcinoma of the colon or rectum that is resistant to available treatment options, including at least two such options from available chemotherapy, targeted and other regimens.
2. Radiographically documented evidence of disease progression from the most recent therapy administered prior to the initiation of BSC.
3. Life expectancy of at least six weeks, in the Investigator's opinion, at the time of disease progression from the most recent therapy administered prior to the initiation of BSC.
4. In the Investigator's opinion, a surgical candidate at the time of disease progression. Initiation of treatment with BSC only within two months.
5. Able to provide written informed consent (by patient or family member or health proxy).

Exclusion Criteria:

Patients who, at the time of disease progression from the most recent therapy administered prior to the initiation of BSC, meet any of the following criteria will be excluded from participating in the study:

1. Documentation of hepatic blood flow abnormalities, i.e., portal vein hypertension and thrombosis, and/or a large volume of ascites.
2. Documentation of concurrent cancer of any other type (Note: patients with non-melanoma skin cancers are still considered eligible).
3. Documentation of positive test result for human immunodeficiency virus (HIV) or any hepatitis (other than Hepatitis A).
4. Considered by the Investigator to be unsuitable for participation in the study upon review of medical history, physical examination or clinical laboratory test results.-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study patient population is composed of patients with treatment-resistant, metastatic colorectal cancer who are only receiving BSC.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Overall Survival | From the date of prior radiographically documented disease progression associated with the most recent therapy administered prior to the initiation of BSC to the date of death, assessed up to 10 years
  Death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Smith, M.D., Ph.D., Study Director — The Rogosin Institute
Locations (1):
- Calvary Hospital, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No